CLINICAL TRIAL: NCT04534647
Title: Serological and Urinary Biomarkers in Latin American Patients With Systemic Lupus Erythematosus: GLADEL 2.0 Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liga Panamericana de Asociaciones de Reumatologia (PANLAR) (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Principal Investigator, Bernardo A Pons-Estel, Clinical Professor, Liga Panamericana de Asociaciones de Reumatologia (PANLAR)
Other Study IDs: GLADEL LUPUS
Record Dates: First submitted 2020-08-24; First posted 2020-09-01 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: different serum and urine biomarkers — urine exosomes and serum biomarkers
  Other Names: Transcriptome studies

SUMMARY:
Lupus nephritis (LN) is one of the main manifestationsin SLE patients, having an important impact on morbidity and mortality. Renal biopsy is the "gold standard" for the diagnosis of LN, however, it is an invasive technique, not free of complications,which is not recommended to be performed serially as a follow-up tool for patients with LN. Searching for biomarkers in SLE has been the subject of interesting research, although results have not always been relevant. Multiple biomarkers have been studied in different locations (soluble markers in blood, urine and biological fluids),of different nature(autoantibodies, genetic markers of "kidney damage") looking atdiagnostic and/orprognostic features. In recent years, several biomarkers have been developed that seek to find an association with pathological patterns, with pathogenic mechanisms and with a non-invasive diagnosis of different glomerulopathies, allowing the identification of prognostic subgroups in each type of kidney disease, while predicting response to treatment and/or recurrence. To date, double-stranded anti-DNA antibodies (anti-dsDNA) and serum complement are the only non-invasive routine biomarkers for monitoring renal activity in patients with LN. However, these markers are only the reflection of the immune activity of the disease and they are not markers of renal damage or poor prognosis. For all the above, the purpose of this study is, in a case-control study, to evaluate simultaneously serum (ANA, anti-dsDNA, anti-C1q, anti-cardiolipin IgG and IgM, anti-ß2GPI IgG and IgM, anti-phosphatidylserine/prothrombin antibodies, and anti-DFS70 antibodies) and urinary biomarkers, and the presence of anti-DFS70 antibodies, in a multiethnic cohort of patients with SLE such as the cohort of GLADEL, and assess its possible correlation with various socio-demographic, clinical and serological manifestations of the disease.

In subgroup of patients, transcriptome studies will be performed using RNA from blood and tissue to identify possible transcriptional signatures.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a diagnosis of SLE will be included. Patients should meet at least one ofthe classification criteria: ACR 1982/1997 (1) and/or SLICC 2012 (2) to determine the efficacy of calcineurin inhibitor-containing treatment regimens in LN cohorts by ethnic groups.
* Age ≥18 years old.
* Patients and controls that volunteer toparticipate and sign the informed consent

Exclusion Criteria:

* Patients with other systemic autoimmune diseases or overlap syndrome (rheumatoid arthritis, systemic sclerosis, dermatomyositis, systemic vasculitis and others).
* Patients who have urinary infection, pregnancy or have a history of hepatitis B, C or HIV virus infection.
* Those patients presenting with antiphospholipid syndrome (APS) associated with lupus will not be excluded from the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Each center will include 25 patients with SLE divided into four groups, each with their corresponding healthy control (ratio 1:1).
  Group 1.Patients with SLE, without renal involvement (never), of any time of disease duration. Total: 10 patients.
  Group 2.Patients with SLE, with prevalent renal involvement (at any time of evolution), currently inactive (*): Total: 5 patients.
  Group 3.Patients with SLE,with prevalent renal involvement (atany time of evolution), currently active (*). Total: 5 patients.
  Group 4.Patients with SLE,with incident renal involvementof recent onset (maximum 3 months), without immunosuppressive treatment and with renal biopsy (mandatory criterion). Total: 5 patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between urinary biomarkers and NL | Baseline to 60 months

SECONDARY OUTCOMES:
Description of clinical features of patients | baseline
Description of immunological characteristics of patients with NL | Baseline to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bernardo Pons-Estel, Rosario, Argentina

IPD SHARING:
Plan to Share IPD: No